CLINICAL TRIAL: NCT06682624
Title: Magnetic Resonance Imaging Pattern Recognition Approach in Pediatric Inherited Neurodegenerative Diseases
Brief Title: MRI in Pediatric Inherited Neurodegnerative Changes
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yasmin Asem Abulelwafa, assisstant lecturer, Sohag University
Other Study IDs: MRI in neurodegenerative
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Neurological Disorder
Keywords: MRI pediatric neurodegenerative diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: MRI — Magnetic Resonance Imaging in recognition of pediatric neurodegenerative disease patterns

SUMMARY:
This study aims to evaluate the diagnostic capability of brain MRI in establishing pattern recognition approach in pediatric inherited neurodegenerative disorders.

Therefore, taking into consideration specific MRI findings, we aim to highlight the potential of MRI to predict the diagnosis of pediatric inherited neurodegenerative diseases.

DETAILED DESCRIPTION:
Pediatric inherited neurodegenerative diseases are non-homogenous group of diseases caused by inborn errors of metabolism (IEMs) that mainly impact the central nervous system. They typically affect newborns and infants . Genetic defects causing specific enzyme deficiencies that lead to deficiency or toxic accumulation of essential metabolites with specific biochemical and molecular abnormalities are the cause of these diseases .

Inborn errors of metabolism are uncommon, which leads to a lack of experience for most neuroradiologists to diagnose these disorders easily. Moreover, most of these disorders manifest in nonspecific manner, creating a diagnostic difficulty for pediatricians, neurologists, and geneticists .

Clinical presentation may be confusing and potentially lead to a delay in the diagnosis and treatment. Incidence of these disorders may vary from one region to another, being higher in communities with consanguineous marriages, ranging from 1.2 to 2 per 100,000 live births. Most exhibit an autosomal recessive mode of inheritance and fewer exhibit an X-linked mode of inheritance.

Multiple methods can be used to classify neurometabolic diseases according to their clinical presentation, biochemical features, impacted cellular organelle, or involved location of the brain.

As a non-invasive means, neuroimaging approaches play a major role in increasing diagnostic accuracy and patient follow-up in IEM by assessing the timing, degree, reversibility, and brain injury.

Imaging based classification includes leukodystrophy (primary involvement of white matter due to genetic abnormality), leukoencephalopathy (secondary involvement of white matter either due to genetic or acquired systemic disorder), poliodystrophy (predominant involvement of grey matter), and pandystrophy (mixed involvement of both white and grey matter).

White matter of the central nervous system is usually affected due to many pathological processes such as delayed myelination (myelin maturation delayed for expected age), hypomyelination (scarcity of myelin or arrest in myelination process), dysmyelination (deposition of abnormally composed fragile myelin), demyelination (secondary loss of myelin that may have been previously normal) and myelinopathy (vacuolation due to deranged brain iron and water hemostasis).

The preferred method for evaluating pediatric inherited neurodegenerative disorders is magnetic resonance imaging (MRI). Examining MRI patterns and clinical indicators aids in narrowing the differential and customizing further laboratory (focused metabolomics) or genetic research.

Magnetic resonance imaging (MRI) can be useful and even crucial for prompt treatment before the receipt of expensive and time-consuming results from genetic or biochemical tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical suspicion of neuro-developmental delay and metabolic disease consulted for or referred to pediatric neurology.
* Patients known to have inherited neurodegenerative diseases under follow-up.

Exclusion Criteria:

- Patients with prior histories of perinatal ischemia or stroke, hypoxic-ischemic encephalopathy, birth trauma or accident, or known systemic diseases (congenital heart disease, renal failure, or autoimmune disorders) will be excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: forty patients of both sexes from day one of life until 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
assessing the MRI patterns of recognition of pediatric neurodegenerative diseases | baseline
  The ability of MRI to diagnose pediatric neurodegenerative diseases based on their characteristic imaging findings correlated to clinical and laboratory findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Knaap MS, Schiffmann R, Mochel F, Wolf NI. Diagnosis, prognosis, and treatment of leukodystrophies. Lancet Neurol. 2019 Oct;18(10):962-972. doi: 10.1016/S1474-4422(19)30143-7. Epub 2019 Jul 12. PMID 31307818
- [Background] Datar R, Prasad AN, Tay KY, Rupar CA, Ohorodnyk P, Miller M, Prasad C. Magnetic resonance imaging in the diagnosis of white matter signal abnormalities. Neuroradiol J. 2018 Aug;31(4):362-371. doi: 10.1177/1971400918764016. Epub 2018 Mar 8. PMID 29517408
- [Background] Loftus JR, Puri S, Meyers SP. Multimodality imaging of neurodegenerative disorders with a focus on multiparametric magnetic resonance and molecular imaging. Insights Imaging. 2023 Jan 16;14(1):8. doi: 10.1186/s13244-022-01358-6. PMID 36645560
- [Background] Lim YT, Mankad K, Kinali M, Tan AP. Neuroimaging Spectrum of Inherited Neurotransmitter Disorders. Neuropediatrics. 2020 Feb;51(1):6-21. doi: 10.1055/s-0039-1698422. Epub 2019 Oct 21. PMID 31634934
- [Background] Lai LM, Gropman AL, Whitehead MT. MR Neuroimaging in Pediatric Inborn Errors of Metabolism. Diagnostics (Basel). 2022 Mar 30;12(4):861. doi: 10.3390/diagnostics12040861. PMID 35453911
- [Background] Alamri A, Aljadhai YI, Alrashed A, Alfheed B, Abdelmoaty R, Alenazi S, Alhashim A, Benini R. Identifying Clinical Clues in Children With Global Developmental Delay / Intellectual Disability With Abnormal Brain Magnetic Resonance Imaging (MRI). J Child Neurol. 2021 May;36(6):432-439. doi: 10.1177/0883073820977330. Epub 2020 Dec 9. PMID 33295251
- [Background] Soni N, Ora M, Bathla G, Nagaraj C, Boles Ponto LL, Graham MM, Saini J, Menda Y. Multiparametric magnetic resonance imaging and positron emission tomography findings in neurodegenerative diseases: Current status and future directions. Neuroradiol J. 2021 Aug;34(4):263-288. doi: 10.1177/1971400921998968. Epub 2021 Mar 5. PMID 33666110
- [Background] Wenger KJ, Koldijk CE, Hattingen E, Porto L, Kurre W. Characterization of MRI White Matter Signal Abnormalities in the Pediatric Population. Children (Basel). 2023 Jan 24;10(2):206. doi: 10.3390/children10020206. PMID 36832335
- [Background] Al Orf A, Waheed KB, Ali EM, Muhammad AK, Al Zahrani FM, Seth SA, Al Jubair NN, Harisi HS, Arulanantham ZJ. Inherited paediatric neurometabolic disorders, can brain magnetic resonance imaging predict? Neurosciences (Riyadh). 2020 Oct;25(5):392-398. doi: 10.17712/nsj.2020.5.20200072. PMID 33459289
- [Background] Aksoy DO, Alkan A. Neurometabolic Diseases in Children: Magnetic Resonance Imaging and Magnetic Resonance Spectroscopy Features. Curr Med Imaging Rev. 2019;15(3):255-268. doi: 10.2174/1573405613666171123152451. PMID 31989877